CLINICAL TRIAL: NCT05733013
Title: Outcomes of Patients With Thyroid Carcinoma Treated With Redifferentiating Agents as Part of Routine Clinical Care: A Prospective Data Collection Study
Brief Title: A Study to Collect Information About the Use of Redifferentiating Medications as a Standard Treatment for Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-320
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Cancer; Thyroid; Refractory Thyroid Cancer
Keywords: RAI refractory thyroid cancer; thyroid cancer; thyroid; Refractory Thyroid Cancer; Radio-iodine refractory thyroid cancer; 22-320; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with refractory thyroid cancer patients
  Interventions: Other: Surveillance Visit

INTERVENTIONS:
Other: Surveillance Visit — Follow-up visits will be carried out at intervals per usual clinical practice. Tolerance of medication and adverse events will be recorded in every visit.

SUMMARY:
The purpose of this study to learn more about the use of redifferentiating medications as a standard treatment for radioactive iodine/RAI-refractory thyroid cancer. This study is a registry study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old at time of consent

Inclusion Criteria:

* Patients diagnosed with RAI refractory thyroid cancer or unlikely to respond to RAI.
* Patients who will receive redifferentiation agents prior to planned diagnostic and/or therapeutic use of radioactive iodine as part of routine clinical care.
* Patients who have never received redifferentiation agents outside of a clinical trial or have received redifferentiation agents in the context of a clinical trial will be enrolled after the clinical team has decided to proceed with a redifferentiation agent as part of routine clinical care prior to diagnostic and/or therapeutic radioactive iodine administration.
* Patients previously treated with redifferentiation agents as part of clinical care prior to diagnostic and/or therapeutic radioactive iodine administration who are willing to provide retrospectively collected data surrounding the time of the previous treatment and will provide prospective data from the time of consent.

Exclusion Criteria:

* RAI refractory thyroid cancer patients that will receive redifferentiation agents prior to diagnostic and/or therapeutic use of radioactive iodine as part of a prospective clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible to receive a redifferentiating agent in the adjuvant setting or in the treatment of structural metastatic disease not enrolled in a clinical trial will be approached for recruitment. All eligible patients will enroll in the study and will be followed indefinitely after enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2028-02-07 (Estimated); Study Completion 2028-02-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events will be collected in every visit | 2 years
  The primary objective of this protocol is to prospectively collect data on patients with radio-iodine refractory thyroid cancer or patients unlikely to respond to radioactive iodine prior, during and after initiation of redifferentiating agents used as part of routine clinical care with or without radioactive iodine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Boucai, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org